CLINICAL TRIAL: NCT03375320
Title: Randomized, Double-Blinded Phase III Study of CABozantinib Versus Placebo IN Patients With Advanced NEuroendocrine Tumors After Progression on Prior Therapy (CABINET)
Brief Title: Testing Cabozantinib in Patients With Advanced Pancreatic Neuroendocrine and Carcinoid Tumors
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2017-02297; NCI-2017-02297 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A021602 (Other: Alliance for Clinical Trials in Oncology); A021602 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2017-12-15; First posted 2017-12-18 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Functioning Pancreatic Neuroendocrine Tumor; Intermediate Grade Lung Neuroendocrine Neoplasm; Locally Advanced Digestive System Neuroendocrine Neoplasm; Locally Advanced Digestive System Neuroendocrine Tumor G1; Locally Advanced Lung Neuroendocrine Neoplasm; Locally Advanced Pancreatic Neuroendocrine Tumor; Locally Advanced Unresectable Digestive System Neuroendocrine Neoplasm; Low Grade Lung Neuroendocrine Neoplasm; Lung Neuroendocrine Tumor; Lung Neuroendocrine Tumor G2; Metastatic Digestive System Neuroendocrine Neoplasm; Metastatic Digestive System Neuroendocrine Tumor G1; Metastatic Lung Neuroendocrine Neoplasm; Metastatic Lung Neuroendocrine Tumor; Metastatic Pancreatic Neuroendocrine Neoplasm; Metastatic Pancreatic Neuroendocrine Tumor; Metastatic Thymus Neuroendocrine Neoplasm; Neuroendocrine Neoplasm; Neuroendocrine Tumor; Neuroendocrine Tumor G2; Non-Functioning Pancreatic Neuroendocrine Tumor; Pancreatic Serotonin-Producing Neuroendocrine Tumor; Thymus Neuroendocrine Tumor; Unresectable Digestive System Neuroendocrine Neoplasm; Unresectable Digestive System Neuroendocrine Tumor G1; Unresectable Lung Neuroendocrine Neoplasm; Unresectable Pancreatic Neuroendocrine Neoplasm; Unresectable Thymus Neuroendocrine Neoplasm
MeSH Terms: conditions — Adenoma, Islet Cell; Neuroendocrine Tumors; Non functioning pancreatic endocrine tumor | interventions — Specimen Handling; cabozantinib; Magnetic Resonance Spectroscopy; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (cabozantinib S-malate) (Experimental): Patients receive cabozantinib S-malate PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood and urine sample collection, and CT, MRI, and/or x-ray imaging during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Procedure: X-Ray Imaging
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood and urine sample collection, and CT, MRI, and/or x-ray imaging during screening and on study. Patients may crossover to receive cabozantinib S-malate at the time of disease progression.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Placebo Administration; Other: Quality-of-Life Assessment; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
  Arms: Arm I (cabozantinib S-malate)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: X-Ray Imaging — Undergo x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase III trial studies cabozantinib to see how well it works compared with placebo in treating patients with neuroendocrine or carcinoid tumors that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). Cabozantinib is a chemotherapy drug known as a tyrosine kinase inhibitor, and it targets specific tyrosine kinase receptors, that when blocked, may slow tumor growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether cabozantinib (cabozantinib S-malate) can significantly improve progression-free survival (PFS) compared to placebo in patients with advanced pancreatic neuroendocrine tumors (NET) whose disease has progressed after prior therapy.

II. To determine whether cabozantinib can significantly improve progression-free survival (PFS) compared to placebo in patients with advanced carcinoid tumors whose disease has progressed after prior therapy.

SECONDARY OBJECTIVES:

I. To determine whether cabozantinib can significantly improve overall survival (OS) compared to placebo in patients with advanced pancreatic NET whose disease has progressed after prior therapy.

II. To determine whether cabozantinib can significantly improve overall survival (OS) compared to placebo in patients with advanced carcinoid tumors whose disease has progressed after prior therapy.

III. To evaluate safety and tolerability of cabozantinib versus placebo in patients with advanced pancreatic NET using Common Terminology Criteria for Adverse Events (CTCAE) and Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).

IV. To evaluate safety and tolerability of cabozantinib versus placebo in patients with advanced carcinoid tumors using CTCAE and PRO-CTCAE.

V. To evaluate the overall radiographic response rate of cabozantinib versus placebo in patients with advanced pancreatic NET whose disease has progressed after prior therapy.

VI. To evaluate the overall radiographic response rate of cabozantinib versus placebo in patients with advanced carcinoid tumors whose disease has progressed after prior therapy.

OTHER OBJECTIVE:

I. Results of the primary analysis will be examined for consistency, while taking into account the stratification factors and/or covariates of baseline quality of life (QOL) and fatigue.

QUALITY OF LIFE SUBSTUDY OBJECTIVE:

I. To compare overall quality of life, disease-related symptoms, and other domains between the two treatment groups (cabozantinib versus [vs.] placebo) within each cohort of patients (pancreatic NET vs. carcinoid tumor). (Quality of Life Substudy Objective - A021602-HO1)

POPULATION PHARMACOKINETICS SUBSTUDY OBJECTIVE:

I. To describe the population pharmacokinetic and exposure-response relationships of cabozantinib in patients with advanced neuroendocrine tumors. (Population Pharmacokinetics Substudy Objective - A021602-PP1)

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive cabozantinib S-malate orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood and urine sample collection, and computed tomography (CT), magnetic resonance imaging (MRI), and/or x-ray imaging during screening and on study.

ARM II: Patients receive placebo PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood and urine sample collection, and CT, MRI, and/or x-ray imaging during screening and on study. Patients may crossover to receive cabozantinib S-malate at the time of disease progression.

After completion of study treatment, patients are followed up every 12 weeks until disease progression or start of new anticancer therapy, and then every 6 months until 8 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of Disease:

  * Histologic Documentation: Well- or moderately-differentiated neuroendocrine tumors of pancreatic and non-pancreatic (i.e. carcinoid) origin by local pathology

    * The pathology report must state ONE of the following: 1) well- or moderately-differentiated neuroendocrine tumor, 2) low- or intermediate-grade neuroendocrine tumor, or 3) carcinoid tumor or atypical carcinoid tumor; documentation of histology from a primary or metastatic site is allowed
    * Patients with poorly differentiated neuroendocrine carcinoma, high-grade neuroendocrine carcinoma without specification of differentiation status, adenocarcinoid tumor, or goblet cell carcinoid tumor are not eligible. Patients with well-differentiated grade 3 neuroendocrine tumor are eligible
  * Stage: Locally advanced/unresectable or metastatic disease
  * Tumor Site: Histological documentation of neuroendocrine tumor of pancreatic, gastrointestinal (GI), lung, thymus, other, or unknown primary site; GI, lung, thymus, other, and unknown primary NETs will enroll in the carcinoid tumor cohort of the study

    * Functional (i.e., associated with symptoms or clinical syndrome related to hormone secretion by tumor) or nonfunctional tumors are allowed
  * Radiologic Evaluation: Target lesions must have shown evidence of disease progression by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria in the 12 months prior to registration; the radiologic images, imaging reports, and clinic notes indicating growth of existing lesions, development of new lesions, or treatment changes must be submitted
* Measurable Disease

  * Patients must have measurable disease per RECIST 1.1 by computer tomography (CT) scan or magnetic resonance imaging (MRI)
  * Lesions must be accurately measured in at least one dimension (longest diameter to be recorded) as >= 1 cm with CT or MRI (or >= 1.5 cm for lymph nodes); non-measurable disease includes disease smaller than these dimensions or lesions considered truly non-measurable including: leptomeningeal disease, ascites, pleural or pericardial effusion, lymphangitic involvement of skin or lung
* Prior Treatment

  * Patient must have experienced disease progression after receiving or intolerance leading to treatment discontinuation of at least one Food and Drug Administration (FDA)-approved line of therapy (except somatostatin analogs); prior lines of therapy must include one of the following: everolimus, sunitinib, or lutetium Lu 177 dotatate in patients with pancreatic NET; everolimus in patients with lung NET; everolimus or lutetium Lu 177 dotatate in patients with gastrointestinal NET
  * Prior treatment (except somatostatin analogs) with biologic therapy, immunotherapy, chemotherapy, investigational agent for malignancy, and/or radiation must be completed at least 28 days prior to registration
  * Prior treatment with somatostatin analogs is allowed, and continuation of treatment with somatostatin analogs while on cabozantinib/placebo is allowed provided that the patient has been on a stable dose for at least two months
  * Prior systemic treatment with radionuclide therapy must be completed at least 6 weeks prior to registration
  * Prior treatment with hepatic artery embolization (including bland embolization, chemoembolization, and selective internal radiation therapy) or ablative therapies is allowed if measurable disease remains outside of the treated area or if there is documented disease progression in a treated site; prior liver-directed or other ablative treatment must be completed at least 28 days prior to registration
  * Prior treatment with cabozantinib is not allowed
  * Patients should have resolution of any toxic effects of prior therapy (except alopecia and fatigue) to National Cancer Institute (NCI) CTCAE, version 5.0, grade 1 or less
  * Patients must have completed any major surgery at least 12 weeks prior to registration and any minor surgery (including uncomplicated tooth extractions) at least 28 days prior to registration; complete wound healing from major surgery must have occurred at least 28 days prior to registration, and complete wound healing from minor surgery must have occurred at least 10 days prior to registration
* Patient History

  * No class III or IV congestive heart failure (CHF) within 6 months of registration
  * No clinically significant cardiac arrhythmia within 6 months of registration
  * No unstable angina or myocardial infarction (MI) within 6 months of registration
  * No thromboembolic events within 6 months of registration (including [incl.] stroke, transient ischemic attack [TIA], deep vein thrombosis [DVT], & pulmonary embolism [PE])
  * No known history of congenital long QT syndrome
  * No uncontrolled hypertension within 14 days of registration (defined as systolic blood pressure [SBP] >= 150 mmHg and/or diastolic blood pressure [DBP] >= 90 mmHg despite optimal medical management)
  * No clinically significant GI bleeding within 6 months of registration
  * No clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding within 6 months of registration including, but not limited to: active peptic ulcer, known endoluminal metastatic lesion(s) with history of bleeding, inflammatory bowel disease, or other gastrointestinal conditions with increased risk of perforation
  * No GI perforation within 6 months of registration
  * No known tumor with invasion into the GI tract from the outside causing increased risk of perforation or bleeding within 28 days of registration
  * No radiologic or clinical evidence of pancreatitis
  * No known cavitary lung lesions
  * No known endobronchial lesions involving the main or lobar bronchi and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage; (CT with contrast is recommended to evaluate such lesions)
  * No hemoptysis greater than 1/2 teaspoon (2.5 mL) or any other signs of pulmonary hemorrhage within the 3 months prior to registration
  * No known tumor invading or encasing any major blood vessels
  * No history of non-healing wounds or ulcers within 28 days of registration
  * No history of fracture within 28 days of registration
  * No brain metastases or cranial epidural disease unless adequately treated, stable, and off steroid support for at least 4 weeks prior to registration
  * No known medical condition causing an inability to swallow oral formulations of agents
  * No history of allergic reaction attributed to compounds of similar chemical or biological composition to cabozantinib/placebo
  * No "currently active" second malignancy other than non-melanoma skin cancers or cervical carcinoma in situ; patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for >= 3 years
* Concomitant Medications

  * Other planned concurrent investigational agents or other tumor directed therapies (chemotherapy, radiation) are not allowed while on this study
  * Concurrent use of somatostatin analogs while on cabozantinib/placebo is allowed provided that the patient has been on a stable dose for at least two months
  * Full dose oral anticoagulation/antiplatelet therapy is not permitted; low dose aspirin =< 81 mg/day is allowed; anticoagulation with therapeutic doses of low molecular weight heparin (LMWH) is allowed in patients who are on a stable dose of LMWH for at least 6 weeks prior to registration; treatment with warfarin is not allowed; anticoagulation in patients with brain metastases is not permitted
  * Chronic concomitant treatment with strong inhibitors of CYP3A4 is not allowed; patients must discontinue the drug at least 14 days prior to registration on the study
  * Chronic concomitant treatment with strong CYP3A4 inducers is not allowed; patients must discontinue the drug at least 14 days prior to registration on the study
* Not pregnant and not nursing

  * Women of childbearing potential must have a negative pregnancy test done =< 14 days prior to registration
  * A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (i.e. has had menses at any time in the preceding 12 consecutive months)
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status: 0-2
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Hemoglobin >= 9 g/dL
* Platelet count >= 100,000/mm^3
* Prothrombin time (PT)/ international normalized ratio (INR), partial thromboplastin time (PTT) < 1.3 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) =< 3 x ULN
* Total bilirubin =< 1.5 x ULN

  * Except in the case of Gilbert disease, in which case total bilirubin must be =< 3 x ULN
* Creatinine =< 1.5 mg/dL OR creatinine clearance >= 45 mL/min
* Albumin >= 2.8 g/dL
* Potassium within normal limits (WNL)

  * Supplementation is acceptable to achieve a value WNL; in patients with low albumin levels, a corrected calcium value WNL is acceptable; in patients with abnormal thyroid stimulating hormone (TSH), if free T4 is normal and patient is clinically euthyroid, patient is eligible
* Phosphorus WNL

  * Supplementation is acceptable to achieve a value WNL; in patients with low albumin levels, a corrected calcium value WNL is acceptable; in patients with abnormal TSH, if free T4 is normal and patient is clinically euthyroid, patient is eligible
* Calcium WNL

  * Supplementation is acceptable to achieve a value WNL; in patients with low albumin levels, a corrected calcium value WNL is acceptable; in patients with abnormal TSH, if free T4 is normal and patient is clinically euthyroid, patient is eligible
* Magnesium WNL

  * Supplementation is acceptable to achieve a value WNL; in patients with low albumin levels, a corrected calcium value WNL is acceptable; in patients with abnormal TSH, if free T4 is normal and patient is clinically euthyroid, patient is eligible
* Urine protein to creatinine (UPC) ratio =< 1
* QT interval corrected for heart rate using Fridericia's formula (QTcF) =< 500 msec
* TSH WNL

  * Supplementation is acceptable to achieve a value WNL; in patients with low albumin levels, a corrected calcium value WNL is acceptable; in patients with abnormal TSH, if free T4 is normal and patient is clinically euthyroid, patient is eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2026-08-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Chan, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (434):
- United States (434):
  - Katmai Oncology Group, Anchorage, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Mills Health Center, San Mateo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - GenesisCare USA - Aventura FP, Aventura, Florida
  - GenesisCare USA - Aventura, Aventura, Florida
  - GenesisCare USA - Boca Ration FP06, Boca Raton, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Memorial Hospital of South Bend, South Bend, Indiana
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Valley Medical Group - Wayne Multispecialty Practice, Wayne, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Farmington Health Center, Farmington, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Strosberg JR, Zemla T, Geyer S, Pulsipher S, Ou FS, Behr S, Raj N, Vijayvergia N, Dasari A, O'Reilly EM, Meyerhardt JA, Wolin EM, Halfdanarson TR, Chan JA. Cabozantinib for advanced grade 3 neuroendocrine tumors: subgroup analysis of the phase 3 CABINET trial (Alliance A021602). Endocr Relat Cancer. 2026 Jan 24;33(1):e250415. doi: 10.1530/ERC-25-0415. Print 2026 Jan 1. PMID 41524552
- [Derived] Chan JA, Geyer S, Zemla T, Knopp MV, Behr S, Pulsipher S, Ou FS, Dueck AC, Acoba J, Shergill A, Wolin EM, Halfdanarson TR, Konda B, Trikalinos NA, Tawfik B, Raj N, Shaheen S, Vijayvergia N, Dasari A, Strosberg JR, Kohn EC, Kulke MH, O'Reilly EM, Meyerhardt JA. Phase 3 Trial of Cabozantinib to Treat Advanced Neuroendocrine Tumors. N Engl J Med. 2025 Feb 13;392(7):653-665. doi: 10.1056/NEJMoa2403991. Epub 2024 Sep 16. PMID 39282913
- [Derived] Kunz PL. Angiogenesis inhibitors in neuroendocrine tumours: finally coming of age. Lancet Oncol. 2020 Nov;21(11):1395-1397. doi: 10.1016/S1470-2045(20)30560-X. No abstract available. PMID 33152282

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm Ia (Cabozantinib S-malate, Extra-pancreatic NET Cohort [epNET]); Arm Ib (Cabozantinib S-malate, Pancreatic NET Cohort [pNET]): Patients receive cabozantinib S-malate PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, and/or x-ray imaging during screening and on study.>
  > Cabozantinib S-malate: Given PO>
  > Computed Tomography: Undergo CT>
  > Magnetic Resonance Imaging: Undergo MRI>
  > Quality-of-Life Assessment: Ancillary studies>
  > X-Ray Imaging: Undergo x-ray
- Arm IIa (Placebo, Extra-pancreatic NET Cohort [epNET]); Arm IIb (Placebo, Pancreatic NET Cohort [pNET]): Patients receive placebo PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, and/or x-ray imaging during screening and on study. Patients may crossover to receive cabozantinib S-malate at the time of disease progression.>
  > Computed Tomography: Undergo CT>
  > Magnetic Resonance Imaging: Undergo MRI>
  > Placebo Administration: Given PO>
  > Quality-of-Life Assessment: Ancillary studies>
  > X-Ray Imaging: Undergo x-ray
Period: Overall Study
Arm/Group | Arm Ia (Cabozantinib S-malate, Extra-pancreatic NET Cohort [epNET]) | Arm IIa (Placebo, Extra-pancreatic NET Cohort [epNET]) | Arm Ib (Cabozantinib S-malate, Pancreatic NET Cohort [pNET]) | Arm IIb (Placebo, Pancreatic NET Cohort [pNET])
Started | 134 | 69 | 64 | 31
Initiated Treatment | 132 | 67 | 63 | 31
Completed | 21 | 7 | 14 | 2
Not Completed | 113 | 62 | 50 | 29
Not completed — Adverse Event | 34 | 9 | 10 | 0
Not completed — Death | 6 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 4 | 5 | 4
Not completed — Progressive disease | 55 | 41 | 29 | 24
Not completed — Alternative treatment | 6 | 1 | 1 | 0
Not completed — Other disease | 1 | 1 | 3 | 0
Not completed — Withdrawal prior to initiation | 2 | 2 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 1 | 1
Not completed — Non-compliance | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm Ia (Cabozantinib S-malate, Extra-pancreatic NET Cohort [epNET]) | Arm IIa (Placebo, Extra-pancreatic NET Cohort [epNET]) | Arm Ib (Cabozantinib S-malate, Pancreatic NET Cohort [pNET]) | Arm IIb (Placebo, Pancreatic NET Cohort [pNET]) | Total
Number analyzed (Participants) | 134 | 69 | 64 | 31 | 298
Age, Continuous [Median (Full Range); unit: years] | 66 [28 to 86] | 66 [30 to 82] | 59.5 [29 to 79] | 64 [39 to 79] | 66 [28 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 31 | 27 | 13 | 145
  Male | 60 | 38 | 37 | 18 | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 2 | 2 | 21
  Not Hispanic or Latino | 125 | 56 | 61 | 26 | 268
  Unknown or Not Reported | 1 | 4 | 1 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 3 | 1 | 4 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 9 | 7 | 3 | 3 | 22
  White | 115 | 55 | 54 | 25 | 249
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 7 | 6 | 0 | 3 | 16
Region of Enrollment [Number; unit: participants]
  United States | 134 | 69 | 64 | 31 | 298

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Will be assessed per Response Evaluation Criteria in Solid Tumors 1.1 determined by retrospective independent central review. Will be compared between treatment arms using the stratified log rank test at one-sided level 0.025. The stratification factors will be used for the analysis. The hazard ratio (HR) for PFS will be estimated using a stratified Cox proportional hazards model, and the 95% confidence interval (CI) for the HR will be provided. Results from an unstratified analysis will also be provided. Kaplan-Meier methodology will be used to estimate the median PFS for each treatment arm, and Kaplan-Meier curves will be produced. Brookmeyer Crowley methodology will be used to construct the 95% CI for the median PFS for each treatment arm.
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm Ia (Cabozantinib S-malate, Extra-pancreatic NET Cohort [epNET]); Arm Ib (Cabozantinib S-malate, Pancreatic NET Cohort [pNET]): Patients receive cabozantinib S-malate PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, and/or x-ray imaging during screening and on study.
  >
  > Cabozantinib S-malate: Given PO
  >
  > Computed Tomography: Undergo CT
  >
  > Magnetic Resonance Imaging: Undergo MRI
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > X-Ray Imaging: Undergo x-ray
- Arm IIa (Placebo, Extra-pancreatic NET Cohort [epNET]); Arm IIb (Placebo, Pancreatic NET Cohort [pNET]): Patients receive placebo PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, and/or x-ray imaging during screening and on study. Patients may crossover to receive cabozantinib S-malate at the time of disease progression.
  >
  > Computed Tomography: Undergo CT
  >
  > Magnetic Resonance Imaging: Undergo MRI
  >
  > Placebo Administration: Given PO
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > X-Ray Imaging: Undergo x-ray
Arm/Group | Arm Ia (Cabozantinib S-malate, Extra-pancreatic NET Cohort [epNET]) | Arm IIa (Placebo, Extra-pancreatic NET Cohort [epNET]) | Arm Ib (Cabozantinib S-malate, Pancreatic NET Cohort [pNET]) | Arm IIb (Placebo, Pancreatic NET Cohort [pNET])
Number analyzed (Participants) | 134 | 69 | 64 | 31
months | 8.4 [7.6 to 12.7] | 3.9 [3.0 to 5.7] | 13.8 [9.2 to 18.5] | 4.4 [3.0 to 5.9]
Statistical Analysis 1: Comparison: Arm Ia (Cabozantinib S-malate, Extra-pancreatic NET Cohort [epNET]) vs Arm IIa (Placebo, Extra-pancreatic NET Cohort [epNET]); Test type: Superiority; p < 0.0001, One-sided unstratified log-rank
Statistical Analysis 2: Comparison: Arm Ib (Cabozantinib S-malate, Pancreatic NET Cohort [pNET]) vs Arm IIb (Placebo, Pancreatic NET Cohort [pNET]); Test type: Superiority; p < 0.0001, One-sided unstratified log-rank

2. Secondary Outcome: Overall Survival (OS)
Description: The analyses for OS will follow intent-to-treat (ITT) principle and will be conducted separately within each cohort (pancreatic neuroendocrine tumor [NET] and carcinoid tumor). The distribution of OS will be estimated using the method of Kaplan-Meier. The median OS, along with the 95% CI, will be estimated by the two treatment groups. Overall survival will be compared between treatment arms using the stratified log-rank test at a one-sided cumulative 2.5% level of significance. The stratified Cox regression will be used to estimate the HR of OS, along with the 95% CI. A hierarchical approach will be used to control for family-wise type-I error rate, therefore OS will be formally statistically tested only if the primary efficacy endpoint, PFS, is statistically significantly different between the two treatment groups.
Time Frame: 60 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm Ia (Cabozantinib S-malate, Extra-pancreatic NET Cohort [epNET]) | Arm IIa (Placebo, Extra-pancreatic NET Cohort [epNET]) | Arm Ib (Cabozantinib S-malate, Pancreatic NET Cohort [pNET]) | Arm IIb (Placebo, Pancreatic NET Cohort [pNET])
Number analyzed (Participants) | 134 | 69 | 64 | 31
months | 21.9 [18.8 to 30.4] | 19.7 [14.2 to 30.0] | 40.0 [31.3 to NA] — Upper end of the confidence interval is not able to be estimated due to a low number of events | 31.1 [23.4 to NA] — Upper end of the confidence interval is not able to be estimated due to a low number of events
Statistical Analysis 1: Comparison: Arm Ia (Cabozantinib S-malate, Extra-pancreatic NET Cohort [epNET]) vs Arm IIa (Placebo, Extra-pancreatic NET Cohort [epNET]); Test type: Superiority; p = 0.2438, One-sided stratified log-rank
Statistical Analysis 2: Comparison: Arm Ib (Cabozantinib S-malate, Pancreatic NET Cohort [pNET]) vs Arm IIb (Placebo, Pancreatic NET Cohort [pNET]); Test type: Superiority; p = 0.4426, One-sided stratified log-rank

3. Secondary Outcome: Number of Patients Experiencing Grade 3+ Adverse Events (AEs) Graded According to the Common Terminology Criteria for Adverse Events (CTCAE) and Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: For CTCAE data, the frequency tables will be reviewed to determine the patterns. The overall adverse event rates will be compared between treatment groups using Chi-square test (or Fisher's exact test if the data in contingency table is sparse). PRO-CTCAE data will, at minimum, be analyzed similarly to CTCAE data. The initial analysis of each PRO-CTCAE item will use all available scores in an analysis which mirrors the approach used for the CTCAE data. Supplemental analysis will use model-based multiple imputation incorporating baseline patient characteristics and physician-rated performance status. CTCAE data may be incorporated as auxiliary data into multiple imputation models for AEs which are captured by both PRO-CTCAE and CTCAE. Results from supplemental analysis will be descriptively compared to the results of the initial analysis to assess the robustness of results to missing data. Additional analyses of PRO-CTCAE data beyond those specified above may be undertaken.
Time Frame: 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm Ia (Cabozantinib S-malate, Extra-pancreatic NET Cohort [epNET]) | Arm IIa (Placebo, Extra-pancreatic NET Cohort [epNET]) | Arm Ib (Cabozantinib S-malate, Pancreatic NET Cohort [pNET]) | Arm IIb (Placebo, Pancreatic NET Cohort [pNET])
Number analyzed (Participants) | 134 | 69 | 64 | 31
Participants | 104 | 47 | 49 | 22

4. Secondary Outcome: Radiographic Response Rate
Description: Will be defined as the proportion of patients in each arm whose best response is either complete response (CR) or partial response (PR). Radiographic response rate for both cohorts: the analyses for confirmed radiographic response rate will follow the ITT principle and will be conducted separately within each cohort (pancreatic NET and carcinoid tumor). The proportion of patients with either confirmed CR or confirmed PR as their best response will be estimated using point estimates and 95% confidence intervals. Radiographic response rate will be compared between treatment arms using the 2-sample z-test to compare sample proportion at a one-sided 2.5% level of significance.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm Ia (Cabozantinib S-malate, Extra-pancreatic NET Cohort [epNET]) | Arm IIa (Placebo, Extra-pancreatic NET Cohort [epNET]) | Arm Ib (Cabozantinib S-malate, Pancreatic NET Cohort [pNET]) | Arm IIb (Placebo, Pancreatic NET Cohort [pNET])
Number analyzed (Participants) | 134 | 69 | 64 | 31
Participants | 7 | 0 | 12 | 0
Statistical Analysis 1: Comparison: Arm Ia (Cabozantinib S-malate, Extra-pancreatic NET Cohort [epNET]) vs Arm IIa (Placebo, Extra-pancreatic NET Cohort [epNET]); Test type: Superiority; p = 0.05, Chi-squared
Statistical Analysis 2: Comparison: Arm Ib (Cabozantinib S-malate, Pancreatic NET Cohort [pNET]) vs Arm IIb (Placebo, Pancreatic NET Cohort [pNET]); Test type: Superiority; p = 0.01, Chi-squared

ADVERSE EVENTS:
Time Frame: 60 months
Groups:
- Arm Ia (Cabozantinib S-malate, Extra-pancreatic NET Cohort [epNET]); Arm Ib (Cabozantinib S-malate, Pancreatic NET Cohort [pNET]): Patients receive cabozantinib S-malate PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, and/or x-ray imaging during screening and on study. >
  * Cabozantinib S-malate: Given PO >
  * Computed Tomography: Undergo CT >
  * Magnetic Resonance Imaging: Undergo MRI >
  * Quality-of-Life Assessment: Ancillary studies >
  * X-Ray Imaging: Undergo x-ray
- Arm IIa (Placebo, Extra-pancreatic NET Cohort [epNET]); Arm IIb (Placebo, Pancreatic NET Cohort [pNET]): Patients receive placebo PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, and/or x-ray imaging during screening and on study. Patients may crossover to receive cabozantinib S-malate at the time of disease progression. >
  * Computed Tomography: Undergo CT >
  * Magnetic Resonance Imaging: Undergo MRI >
  * Placebo Administration: Given PO >
  * Quality-of-Life Assessment: Ancillary studies >
  * X-Ray Imaging: Undergo x-ray
Arm/Group | Arm Ia (Cabozantinib S-malate, Extra-pancreatic NET Cohort [epNET]) | Arm IIa (Placebo, Extra-pancreatic NET Cohort [epNET]) | Arm Ib (Cabozantinib S-malate, Pancreatic NET Cohort [pNET]) | Arm IIb (Placebo, Pancreatic NET Cohort [pNET])
All-Cause Mortality (participants affected / at risk) | 60/134 | 37/69 | 21/64 | 11/31
Serious Adverse Events (participants affected / at risk) | 89/134 | 41/69 | 49/64 | 21/31
Other Adverse Events (participants affected / at risk) | 134/134 | 69/69 | 64/64 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm Ia (Cabozantinib S-malate, Extra-pancreatic NET Cohort [epNET]) (N=134) | Arm IIa (Placebo, Extra-pancreatic NET Cohort [epNET]) (N=69) | Arm Ib (Cabozantinib S-malate, Pancreatic NET Cohort [pNET]) (N=64) | Arm IIb (Placebo, Pancreatic NET Cohort [pNET]) (N=31)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 5 (5) | 4 (4) | 4 (4)
Acute intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 2 (3) | 1 (1) | 2 (2)
Acute Metabolic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Alkaline phosphatase increased (Investigations) | 5 (5) | 4 (4) | 2 (2) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial thromboembolism (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (4) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Atrial defect (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Bacteremia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 6 (6) | 3 (3) | 3 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 1 (4) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Craniotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cushing's Syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death NOS (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 15 (15) | 5 (5) | 4 (4) | 0 (0)
Disease progression (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 2 (14) | 0 (0) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exploratory laparotomy; enterectomy with anastomosis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 15 (15) | 7 (7) | 10 (10) | 4 (4)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (9) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
GGT increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (7) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 5 (5) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (19) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 30 (30) | 5 (5) | 16 (16) | 8 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 4 (5) | 0 (0)
Intrahepatic biliary dilation (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Large Bowel Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 13 (13) | 1 (1) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MRSE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 4 (4) | 1 (1) | 5 (5) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 5 (5) | 2 (2)
Neuroendocrine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (12)
Pain (General disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 5 (5) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (7) | 0 (0)
Reversbl posterior leukoenceph syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right foot drop (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salmonella Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Severe LAD occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (4) | 1 (1) | 1 (2) | 3 (5)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spontaneous bacterial peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Strangulated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subendocardial ischemia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sudden death NOS (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 5 (6) | 4 (4) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 2 (2) | 8 (8) | 0 (0)
Tooth Extraction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureter Perforation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2) | 4 (4) | 2 (2)
Weight loss (Investigations) | 6 (6) | 1 (1) | 2 (2) | 1 (1)
White blood cell decreased (Investigations) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm Ia (Cabozantinib S-malate, Extra-pancreatic NET Cohort [epNET]) (N=134) | Arm IIa (Placebo, Extra-pancreatic NET Cohort [epNET]) (N=69) | Arm Ib (Cabozantinib S-malate, Pancreatic NET Cohort [pNET]) (N=64) | Arm IIb (Placebo, Pancreatic NET Cohort [pNET]) (N=31)
Abdominal distension (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (9) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 34 (159) | 22 (48) | 13 (75) | 3 (14)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial throm time prolonged (Investigations) | 0 (0) | 0 (0) | 2 (20) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 89 (455) | 15 (31) | 49 (355) | 12 (29)
Alkaline phosphatase increased (Investigations) | 38 (186) | 17 (50) | 14 (98) | 9 (32)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 11 (62) | 0 (0) | 3 (24) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (93) | 0 (0) | 7 (72) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (21) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Anal pain (Gastrointestinal disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 44 (256) | 17 (63) | 18 (113) | 9 (38)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 47 (262) | 9 (28) | 14 (80) | 5 (14)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 12 (103) | 3 (24) | 6 (43) | 4 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (20) | 2 (2) | 7 (31) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 6 (45) | 1 (21) | 2 (6) | 1 (4)
Ascites (Gastrointestinal disorders) | 3 (17) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 96 (595) | 17 (38) | 50 (370) | 15 (30)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (104) | 10 (32) | 8 (38) | 4 (8)
Belching (Gastrointestinal disorders) | 2 (6) | 0 (0) | 2 (7) | 0 (0)
Biliary fistula (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 10 (66) | 3 (12) | 4 (45) | 0 (0)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 1 (5) | 0 (0)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 20 (72) | 5 (9) | 8 (13) | 1 (3)
Blood lactate dehydrogenase increased (Investigations) | 9 (102) | 0 (0) | 4 (43) | 0 (0)
Blurred vision (Eye disorders) | 6 (31) | 3 (5) | 4 (35) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (49) | 3 (12) | 1 (37) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 4 (29) | 0 (0) | 4 (52) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 4 (22) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 5 (53) | 2 (17) | 1 (1) | 1 (4)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 2 (9) | 0 (0)
Cataract (Eye disorders) | 1 (13) | 0 (0) | 1 (2) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 8 (15) | 1 (1) | 2 (2) | 2 (2)
Cholesterol high (Investigations) | 1 (1) | 1 (8) | 3 (20) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 2 (17) | 0 (0) | 2 (26) | 1 (3)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Confusion (Psychiatric disorders) | 3 (7) | 1 (3) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 22 (122) | 9 (30) | 8 (63) | 8 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (77) | 7 (9) | 10 (20) | 1 (4)
Creatinine increased (Investigations) | 31 (124) | 9 (21) | 5 (48) | 6 (9)
Dehydration (Metabolism and nutrition disorders) | 12 (18) | 2 (4) | 5 (8) | 2 (4)
Delusions (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 12 (90) | 5 (39) | 0 (0) | 3 (9)
Diarrhea (Gastrointestinal disorders) | 82 (773) | 31 (145) | 40 (369) | 10 (28)
Dizziness (Nervous system disorders) | 22 (60) | 4 (9) | 16 (32) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (15) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 21 (163) | 5 (24) | 3 (30) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (111) | 3 (12) | 7 (26) | 2 (13)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysesthesia (Nervous system disorders) | 4 (19) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 49 (339) | 1 (2) | 20 (153) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (11) | 1 (3) | 3 (11) | 1 (3)
Dysphagia (Gastrointestinal disorders) | 4 (8) | 1 (1) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 (101) | 9 (21) | 12 (51) | 2 (5)
Dysuria (painful urination) (Renal and urinary disorders) | 2 (10) | 3 (5) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 4 (26) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 2 (5) | 1 (3) | 0 (0)
ECG QT corrected interval prolonged (Investigations) | 4 (6) | 0 (0) | 3 (4) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 20 (135) | 5 (13) | 4 (12) | 3 (6)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (5) | 0 (0) | 3 (8) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 6 (27) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (57) | 0 (0) | 4 (13) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 8 (34) | 1 (5) | 1 (9) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 8 (13) | 2 (3) | 1 (1) | 0 (0)
Fatigue (General disorders) | 103 (951) | 42 (177) | 48 (492) | 17 (95)
Fecal incontinence (Gastrointestinal disorders) | 2 (17) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 4 (5) | 1 (1) | 4 (26) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (32) | 1 (3) | 3 (31) | 0 (0)
Flatulence (Gastrointestinal disorders) | 14 (103) | 1 (1) | 4 (22) | 0 (0)
Floaters (Eye disorders) | 1 (2) | 0 (0) | 1 (5) | 0 (0)
Flu like symptoms (General disorders) | 3 (6) | 0 (0) | 4 (8) | 0 (0)
Flushing (Vascular disorders) | 16 (127) | 10 (60) | 5 (16) | 1 (4)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 3 (16) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 3 (11) | 0 (0) | 1 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 20 (157) | 3 (9) | 10 (90) | 1 (4)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 8 (49) | 4 (11) | 6 (56) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 3 (19) | 0 (0) | 2 (13) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 2 (2) | 0 (0) | 1 (7) | 0 (0)
Generalized edema (General disorders) | 3 (15) | 1 (2) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 13 (41) | 1 (2) | 0 (0) | 1 (2)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gum infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair color changes (Skin and subcutaneous tissue disorders) | 13 (110) | 0 (0) | 7 (74) | 0 (0)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 2 (18) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 24 (102) | 9 (18) | 10 (75) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 4 (41) | 1 (1) | 1 (4) | 1 (4)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (5) | 1 (2) | 0 (0) | 0 (0)
Hemoglobin increased (Investigations) | 3 (8) | 0 (0) | 1 (2) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 5 (37) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 11 (74) | 2 (2) | 7 (80) | 0 (0)
Hot flashes (Vascular disorders) | 3 (21) | 3 (5) | 1 (20) | 2 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (6) | 5 (5) | 1 (1) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 50 (297) | 25 (128) | 26 (234) | 15 (61)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (17) | 1 (3) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 12 (37) | 6 (8) | 7 (23) | 3 (8)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (7) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidemia (Metabolism and nutrition disorders) | 4 (33) | 2 (4) | 0 (0) | 1 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 6 (9) | 0 (0) | 3 (5) | 3 (15)
Hypernatremia (Metabolism and nutrition disorders) | 2 (17) | 3 (7) | 1 (1) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 3 (12) | 1 (2) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 65 (828) | 27 (148) | 31 (461) | 11 (69)
Hyperthyroidism (Endocrine disorders) | 4 (7) | 0 (0) | 4 (13) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 1 (21) | 1 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 30 (118) | 5 (9) | 11 (48) | 4 (16)
Hypocalcemia (Metabolism and nutrition disorders) | 28 (92) | 4 (5) | 15 (50) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 9 (18) | 1 (3) | 7 (10) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 26 (62) | 5 (21) | 6 (30) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 26 (149) | 2 (16) | 7 (50) | 2 (6)
Hyponatremia (Metabolism and nutrition disorders) | 24 (76) | 4 (8) | 11 (41) | 5 (12)
Hypophosphatemia (Metabolism and nutrition disorders) | 25 (71) | 4 (7) | 16 (69) | 2 (4)
Hypotension (Vascular disorders) | 7 (17) | 0 (0) | 5 (13) | 1 (1)
Hypothyroidism (Endocrine disorders) | 49 (385) | 5 (48) | 21 (242) | 3 (9)
Infections and infestations - Oth spec (Infections and infestations) | 10 (12) | 2 (2) | 6 (6) | 1 (1)
INR increased (Investigations) | 3 (23) | 1 (1) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 11 (52) | 5 (15) | 4 (18) | 1 (2)
Intracranial hemorrhage (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (1) | 1 (2) | 2 (5) | 1 (5)
Joint infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (18) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (8) | 0 (0) | 1 (6) | 1 (2)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Localized edema (General disorders) | 5 (23) | 0 (0) | 2 (24) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 27 (388) | 12 (43) | 12 (82) | 5 (9)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 3 (9) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 2 (7) | 0 (0) | 0 (0) | 1 (3)
Malaise (General disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 3 (7) | 2 (3) | 1 (22) | 0 (0)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (2) | 1 (38) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 48 (239) | 6 (10) | 26 (174) | 2 (3)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 18 (90) | 1 (3) | 10 (48) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 4 (32) | 2 (22) | 3 (44) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (61) | 2 (3) | 5 (37) | 2 (15)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (12) | 1 (1) | 4 (52) | 1 (2)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0) | 1 (3) | 0 (0)
Nail infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (13) | 3 (4) | 1 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 53 (281) | 13 (33) | 21 (126) | 8 (23)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (8) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 3 (32) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (3) | 0 (0) | 2 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 49 (251) | 2 (4) | 17 (93) | 2 (3)
Night blindness (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 11 (17) | 2 (3) | 9 (24) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 8 (41) | 0 (0) | 4 (31) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 4 (10) | 0 (0) | 5 (36) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 15 (47) | 7 (33) | 4 (6) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (66) | 2 (4) | 3 (34) | 1 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 47 (334) | 5 (8) | 24 (247) | 5 (10)
Palpitations (Cardiac disorders) | 0 (0) | 2 (23) | 2 (11) | 0 (0)
Papulopustular rash (Infections and infestations) | 1 (4) | 0 (0) | 1 (7) | 0 (0)
Paresthesia (Nervous system disorders) | 3 (11) | 2 (24) | 5 (32) | 1 (3)
Paronychia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 2 (13) | 1 (2) | 1 (23) | 1 (2)
Penile infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (11) | 0 (0) | 0 (0) | 0 (0)
Periorbital edema (Eye disorders) | 3 (5) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 5 (15) | 0 (0) | 0 (0) | 2 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (90) | 1 (3) | 4 (12) | 3 (5)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 74 (434) | 8 (30) | 24 (149) | 6 (21)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 1 (1) | 1 (4)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (19) | 2 (8) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (9) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (13) | 1 (1) | 2 (4) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Premature menopause (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 2 (20) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (16) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 11 (49) | 3 (6) | 4 (18) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (22) | 2 (5) | 1 (25) | 2 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 37 (141) | 3 (5) | 14 (77) | 4 (6)
Rash pustular (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 4 (16) | 0 (0) | 1 (10) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 0 (0) | 1 (2) | 2 (16) | 2 (10)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (5) | 1 (1) | 0 (0)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 3 (9) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 1 (6) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 2 (10) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 8 (35) | 2 (6) | 3 (23) | 2 (5)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 9 (32) | 2 (3) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 18 (141) | 2 (2) | 6 (30) | 2 (5)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (13) | 0 (0) | 1 (8) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (10) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (3) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6) | 0 (0) | 1 (4)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 8 (37) | 2 (5) | 6 (20) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (4) | 1 (2)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (10) | 1 (3) | 0 (0)
Testicular disorder (Reproductive system and breast disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0) | 4 (41) | 1 (1)
Thrush (Infections and infestations) | 4 (6) | 0 (0) | 2 (8) | 0 (0)
Thyroid stimulating hormone increased (Investigations) | 8 (41) | 2 (4) | 8 (65) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 4 (23) | 4 (32) | 3 (49) | 0 (0)
Tooth discoloration (Gastrointestinal disorders) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 5 (8) | 0 (0) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (24) | 0 (0)
Tremor (Nervous system disorders) | 4 (12) | 0 (0) | 0 (0) | 0 (0)
Tricuspid valve disease (Cardiac disorders) | 1 (10) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (20) | 2 (3) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 6 (7) | 0 (0) | 2 (4) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (3) | 2 (8) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (17) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (25) | 2 (3) | 5 (34) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 3 (5) | 2 (2) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (18) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (10) | 2 (4) | 1 (6) | 0 (0)
Viremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision decreased (Eye disorders) | 2 (16) | 0 (0) | 0 (0) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 (24) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 22 (70) | 5 (8) | 14 (29) | 3 (7)
Watering eyes (Eye disorders) | 1 (9) | 0 (0) | 0 (0) | 0 (0)
Weight gain (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 35 (300) | 3 (4) | 10 (91) | 1 (12)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 45 (311) | 2 (11) | 12 (59) | 1 (2)
Wound complication (Injury, poisoning and procedural complications) | 3 (13) | 0 (0) | 1 (3) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT03375320/Prot_SAP_000.pdf